CLINICAL TRIAL: NCT06305013
Title: Pulseless Electrical Activity: the Ability of Nurses to Recognize It
Brief Title: PEA: the Ability of Nurses to Recognize It (PEA: ANTRI)
Acronym: PEARECOG
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Department of Simulation Medicine, Faculty of Medicine, Masaryk University (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: SIMU PEA 2024
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pulseless Electrical Activity
Keywords: Pulseless electrical activity; recognition; nurse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participant of simulation course organised by Department of Simulation medicine: Participant of simulation course organised by Department of Simulation medicine
  Interventions: Other: Pulseless electrical activity recognition

INTERVENTIONS:
Other: Pulseless electrical activity recognition — The ability of nurses to recognize the pulseless electrical activity in the questionnaire (electronic survey)

SUMMARY:
The Ability to recognize cardiac arrest is crucial in emergency situations and all health care professionals should be able to do so. The identification of pulseless electrical activity can be difficult even if the theoretical knowledge of this state is well known. This research will be performed at the Simulation centre of Medical Faculty, Masaryk university and it will be focused on nurses who will come to the simulation course. All the participants will get prelearning theoretical materials that will contain chapter about pulseless electrical activity and its recognition. In the beginning of the course they will be asked to fill up the questionnaire with four different pictures of patient´s monitor in cardiac arrest. It will be evaluated whether the pulseless electrical activity will be recognized.

DETAILED DESCRIPTION:
The Ability to recognize cardiac arrest is crucial in emergency situations and all health care professionals should be able to do so. The identification of pulseless electrical activity can be difficult even if the theoretical knowledge of this state is well known. This research will be performed at the Simulation centre of Medical Faculty, Masaryk university and it will be focused on nurses who will come to the simulation course. All the participants will get prelearning theoretical materials that will contain chapter about pulseless electrical activity and its recognition. In the beginning of the course they will be asked to fill up the questionnaire with four different pictures of patient´s monitor in cardiac arrest. It will be evaluated whether the pulseless electrical activity will be recognized.

ELIGIBILITY:
Inclusion Criteria:

* Nurse or paramedic
* Participant of simulation course organised by Department of Simulation medicine, Faculty of medicine, Masaryk university

Exclusion Criteria:

* No experience wiht monitoring patients by vital signs monitor

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant of simulation course organised by Department of Simulation medicine, Faculty of medicine, Masaryk university
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Pulseless electrical activity recognition, | 12 months
  The ability of nurses to recognize the pulseless electrical activity in the questionnaire (electronic survey)

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kosinová, assoc. prof, Study Chair — Department of Simulation Medicine, Faculty of Medicine, Masaryk University
Locations (1):
- Faculty hospital Brno, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided